CLINICAL TRIAL: NCT03642769
Title: Lactated Ringer's Versus Normal Saline in the Management of Acute Pancreatitis
Brief Title: Lactated Ringer's Versus Normal Saline for Acute Pancreatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, James Buxbaum, Principal Investigator, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: APP-17-06494
Record Dates: First submitted 2018-02-12; First posted 2018-08-22 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-12

CONDITIONS: Pancreatitis, Acute
Keywords: Pancreatitis; Fluids; SIRS; Management; Lactated Ringer; Normal Saline
MeSH Terms: conditions — Pancreatitis | interventions — Hypodermoclysis; Fluid Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lactated Ringer (Active Comparator): Patients will receive fluid administration of Lactated Ringer's solution at a pre-determined volume algorithm that is the same for both arms
  Interventions: Other: Fluid administration
- Normal Saline (Experimental): Patients will receive fluid administration of Normal Saline solution at a pre-determined volume algorithm that is the same for both arms
  Interventions: Other: Fluid administration

INTERVENTIONS:
Other: Fluid administration — Fluid administration of bolus and maintenance fluids
  Other Names: Fluid

SUMMARY:
Acute pancreatitis is a common problem in the United States necessitating 275,000 hospital admissions per year, with resultant healthcare costs of approximately 2.5 billion USD annually. As numerous trials have failed to show a benefit to specific pharmacologic therapies in acute pancreatitis, the mainstay of treatment has been both supportive care and early, aggressive fluid resuscitation. Small randomized studies have shown conflicting results with regards to the influence of resuscitation fluid on outcomes in acute pancreatitis, necessitating a large randomized trial to clarify if fluid choice matters or not in the treatment of acute pancreatitis.

The objective of this study is to assess the comparative efficacy of normal saline versus lactated ringer's solution in the management of acute pancreatitis.

Patients presenting to the Los Angeles County Hospital with acute pancreatitis will be randomized to fluid resuscitation with NS or LR with volumes of fluid administered according to a pre-determined algorithm that will be the same for both treatment arms.

The primary outcome of the study will be the change in SIRS prevalence from enrollment to 24 hours. Secondary outcomes will include the change in SIRS prevalence from enrollment to 48 hours and 72 hours, development of moderately severe or severe pancreatitis, change in PASS score, ICU admission, length of hospitalization, persistent pain or disability after discharge, and time of advancement to oral diet and discharge.

DETAILED DESCRIPTION:
Background: Acute pancreatitis is a common problem in the United States necessitating 275,000 hospital admissions per year, with resultant healthcare costs of approximately 2.5 billion USD annually. As numerous trials have failed to show a benefit to specific pharmacologic therapies in acute pancreatitis, the mainstay of treatment has been both supportive care and early, aggressive fluid resuscitation. Small randomized studies have shown conflicting results with regards to the influence of resuscitation fluid on outcomes in acute pancreatitis, necessitating a large randomized trial to clarify if fluid choice matters or not in the treatment of acute pancreatitis.

Objective: To assess the comparative efficacy of normal saline versus lactated ringer's solution in the management of acute pancreatitis.

Study Design: Patients presenting to the Los Angeles County Hospital with acute pancreatitis are the focus population of this study. Patients will be randomized to fluid resuscitation with NS or LR within 8 hours of diagnosis of pancreatitis. The inclusion and exclusion criterion will be assessed (see below). Randomization will be performed using a random sequence algorithm with concealed allocation. The patients will be blinded to allocation by covering the bag with an opaque covering. A study physician determining the outcomes will also be blinded. Following randomization, the volumes of fluid administered for the resuscitation will be determined by a pre-determined algorithm that will be the same for both treatment arms. The hydration algorithm is as follows: all patients will receive a bolus of the treatment fluid at a rate of 5 mL/kg/hour to be administered over the first two hours (total 10 mL/kg) with an assessment for volume overload at 1 hour. They will then will receive maintenance fluids at a rate of 3 mL/kg/hour. After 12 hours participants will have blood urea nitrogen (BUN) assessed, which is part of the standard clinical procedure. Those who do not have a fall in this parameter or who develop SIRS by this 12 hour checkpoint will receive a second 5 mL/kg/hour bolus over two hours (as above) of their designated treatment fluid followed by further treatment fluid at a rate of 3 mL/kg/hour. Those who do have a fall in BUN will receive further treatment fluid at a rate of 3 mL/kg/hour for 12 additional hours. Patients' volume status will be assessed in the following manner: study physicians will perform a targeted physical exam which will include assessment of JVD, lung auscultation, and monitoring for edema Q12 hours for the first 24 hours, then daily for the remainder of the hospital admission. In elderly patients and those with co-morbidities, the targeted physical exam will be performed Q12 hours for the entire hospital admission. Vitals will also be obtained Q6-8 hours. If they develop signs of fluid overload including pitting edema, ascites, anasacra, pulmonary edema, or dyspnea, or signs of renal failure including oliguria, anuria, or hypotension, they will have their fluid rate managed at the discretion of their treating physicians. However, it will be requested that if further fluid is given that it be the assigned type (LR versus NS). At 24 hours patients will be assessed for SIRS development (see outcomes). Beyond this point fluid rate will be per the primary team though it still be encouraged that the assigned type of fluid (LR versus NS) is used for additional resuscitation with the rate and volume beyond this point at the discretion of the treating physician. However, if the treating physicians have a strong preference to change to a different fluid type for clinical reasons this will be recorded (for post hoc analysis) and the patient included in the intention to treat analysis.

ELIGIBILITY:
Inclusion Criteria:

* Presentation with acute pancreatitis as defined by two of three criterion; amylase or lipase > 3x the upper limit of normal, classical abdominal pain, or imaging suggestive of pancreatitis. Such radiographic findings include swelling, edema, or heterogeneity of the gland or peripancreatic fluid or stranding.

Exclusion Criteria:

* Patients with severe pancreatitis as defined by the Revised Atlanta Classification will be excluded. Severe pancreatitis is defined by the Revised Atlanta Classification as those with a Modified Marshall score of >2 for their cardiovascular renal, or respiratory system will be excluded (Figure 2).13 Practically this includes patients with systolic blood pressure <90, serum creatinine >1.9, and PaO2/FiO2 <300 (Figure 3). Since blood gases are unlikely to be drawn on those with mild pancreatitis we will exclude patients with an oxygen saturation <92% on room air and certainly any patients which require intubation for respiratory failure due to pancreatitis.
* Patients who cannot tolerate increased doses of fluids for other reasons will also be excluded. This consists of those with cardiac insufficiency (CI, >NYHA Class II heart failure), pulmonary edema, dialysis requirement, or severe liver dysfunction (albumin < 3mg/dL, known cirrhosis).
* Pregnant women will also be excluded as they are prone to retain sodium and water, which puts them at increased risk of pulmonary congestion, ascites or peripheral edema.
* Patients who are incarcerated, younger than eighteen, or unable to give informed consent will be excluded.
* Individuals who present with clinical signs of edema or anasacra, including pulmonary congestion, peripheral swelling, and ascites, will also be ineligible for the study.
* Administration of fluids prior to the enrollment in the study will not be an exclusion criterion as this reflects actual clinical practice (hydration during evaluation period) however all fluids given prior to the study will be meticulously recorded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2018-09-18 (Actual); Primary Completion 2021-08-16 (Actual); Study Completion 2021-08-16 (Actual)

PRIMARY OUTCOMES:
SIRS at 24 hours | 24 hours
  Change in SIRS prevalence from enrollment to 24 hours

SECONDARY OUTCOMES:
SIRS at 48 hours | 48 hours
  Proportion of patients with change in SIRS from enrollment to 48 hours
SIRS at 72 hours | 72 hours
  Change in SIRS prevalence from enrollment to 72 hours
Moderately severe acute pancreatitis | 48 hours
  Development of moderately severe acute pancreatitis
Severe acute pancreatitis | >48 hours
  Development of severe acute pancreatitis
PASS score | 24 hours
  Change in PASS score from enrollment to 24 hours
PASS score | 48 hours
  Change in PASS score from enrollment to 48 hours
PASS score | 72 hours
  Change in PASS score from enrollment to 72 hours
ICU admission | >72 hours
  ICU admission and ICU intervention including intubation, respiratory distress with out intubation defined as RR>20 AND O2 Sat<90% on room air, death, development of extrapancreatic fluid collection (EPFS)
Length of hospitalization | >72 hours
  Length of hospitalization
Pain after discharge based on a 0-10 intensity scale (10 most severe, 0 none) | 2 weeks
  Report of persistent pain or disability after discharge based on telephone follow-up based on a 0-10 intensity scale (10 most severe, 0 none)
Advance diet | >48 hours
  Time to advancement of oral diet
Time to work | 2 weeks
  Time to work after hospitalization based on post-discharge telephone follow-up

CONTACTS AND LOCATIONS:
Overall Officials: James Buxbaum, MD, Principal Investigator — University of Southern California
Locations (1):
- LAC+USC Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tenner S, Baillie J, DeWitt J, Vege SS; American College of Gastroenterology. American College of Gastroenterology guideline: management of acute pancreatitis. Am J Gastroenterol. 2013 Sep;108(9):1400-15; 1416. doi: 10.1038/ajg.2013.218. Epub 2013 Jul 30. PMID 23896955
- [Background] Singh VK, Gardner TB, Papachristou GI, Rey-Riveiro M, Faghih M, Koutroumpakis E, Afghani E, Acevedo-Piedra NG, Seth N, Sinha A, Quesada-Vazquez N, Moya-Hoyo N, Sanchez-Marin C, Martinez J, Lluis F, Whitcomb DC, Zapater P, de-Madaria E. An international multicenter study of early intravenous fluid administration and outcome in acute pancreatitis. United European Gastroenterol J. 2017 Jun;5(4):491-498. doi: 10.1177/2050640616671077. Epub 2016 Sep 20. PMID 28588879
- [Background] Forsmark CE, Vege SS, Wilcox CM. Acute Pancreatitis. N Engl J Med. 2016 Nov 17;375(20):1972-1981. doi: 10.1056/NEJMra1505202. No abstract available. PMID 27959604
- [Background] Buxbaum JL, Quezada M, Da B, Jani N, Lane C, Mwengela D, Kelly T, Jhun P, Dhanireddy K, Laine L. Early Aggressive Hydration Hastens Clinical Improvement in Mild Acute Pancreatitis. Am J Gastroenterol. 2017 May;112(5):797-803. doi: 10.1038/ajg.2017.40. Epub 2017 Mar 7. PMID 28266591
- [Background] Cuthbertson CM, Christophi C. Disturbances of the microcirculation in acute pancreatitis. Br J Surg. 2006 May;93(5):518-30. doi: 10.1002/bjs.5316. PMID 16607683
- [Background] Raghunathan K, Shaw A, Nathanson B, Sturmer T, Brookhart A, Stefan MS, Setoguchi S, Beadles C, Lindenauer PK. Association between the choice of IV crystalloid and in-hospital mortality among critically ill adults with sepsis*. Crit Care Med. 2014 Jul;42(7):1585-91. doi: 10.1097/CCM.0000000000000305. PMID 24674927
- [Background] Rochwerg B, Alhazzani W, Sindi A, Heels-Ansdell D, Thabane L, Fox-Robichaud A, Mbuagbaw L, Szczeklik W, Alshamsi F, Altayyar S, Ip WC, Li G, Wang M, Wludarczyk A, Zhou Q, Guyatt GH, Cook DJ, Jaeschke R, Annane D; Fluids in Sepsis and Septic Shock Group. Fluid resuscitation in sepsis: a systematic review and network meta-analysis. Ann Intern Med. 2014 Sep 2;161(5):347-55. doi: 10.7326/M14-0178. PMID 25047428
- [Background] Correa TD, Cavalcanti AB, Assuncao MS. Balanced crystalloids for septic shock resuscitation. Rev Bras Ter Intensiva. 2016 Oct-Dec;28(4):463-471. doi: 10.5935/0103-507X.20160079. PMID 28099643
- [Background] Wu BU, Hwang JQ, Gardner TH, Repas K, Delee R, Yu S, Smith B, Banks PA, Conwell DL. Lactated Ringer's solution reduces systemic inflammation compared with saline in patients with acute pancreatitis. Clin Gastroenterol Hepatol. 2011 Aug;9(8):710-717.e1. doi: 10.1016/j.cgh.2011.04.026. Epub 2011 May 12. PMID 21645639
- [Background] Lipinski M, Rydzewska-Rosolowska A, Rydzewski A, Rydzewska G. Fluid resuscitation in acute pancreatitis: Normal saline or lactated Ringer's solution? World J Gastroenterol. 2015 Aug 21;21(31):9367-72. doi: 10.3748/wjg.v21.i31.9367. PMID 26309362
- [Background] de-Madaria E, Soler-Sala G, Lopez-Font I, Zapater P, Martinez J, Gomez-Escolar L, Sanchez-Fortun C, Sempere L, Perez-Lopez J, Lluis F, Perez-Mateo M. Update of the Atlanta Classification of severity of acute pancreatitis: should a moderate category be included? Pancreatology. 2010;10(5):613-9. doi: 10.1159/000308795. Epub 2010 Oct 30. PMID 21042037
- [Background] Balthazar EJ. Acute pancreatitis: assessment of severity with clinical and CT evaluation. Radiology. 2002 Jun;223(3):603-13. doi: 10.1148/radiol.2233010680. PMID 12034923
- [Background] Warndorf MG, Kurtzman JT, Bartel MJ, Cox M, Mackenzie T, Robinson S, Burchard PR, Gordon SR, Gardner TB. Early fluid resuscitation reduces morbidity among patients with acute pancreatitis. Clin Gastroenterol Hepatol. 2011 Aug;9(8):705-9. doi: 10.1016/j.cgh.2011.03.032. Epub 2011 Apr 8. PMID 21554987
- [Background] Cotton PB, Lehman G, Vennes J, Geenen JE, Russell RC, Meyers WC, Liguory C, Nickl N. Endoscopic sphincterotomy complications and their management: an attempt at consensus. Gastrointest Endosc. 1991 May-Jun;37(3):383-93. doi: 10.1016/s0016-5107(91)70740-2. PMID 2070995
- [Background] Banks PA, Bollen TL, Dervenis C, Gooszen HG, Johnson CD, Sarr MG, Tsiotos GG, Vege SS; Acute Pancreatitis Classification Working Group. Classification of acute pancreatitis--2012: revision of the Atlanta classification and definitions by international consensus. Gut. 2013 Jan;62(1):102-11. doi: 10.1136/gutjnl-2012-302779. Epub 2012 Oct 25. PMID 23100216
- [Background] Wu BU, Batech M, Quezada M, Lew D, Fujikawa K, Kung J, Jamil LH, Chen W, Afghani E, Reicher S, Buxbaum J, Pandol SJ. Dynamic Measurement of Disease Activity in Acute Pancreatitis: The Pancreatitis Activity Scoring System. Am J Gastroenterol. 2017 Jul;112(7):1144-1152. doi: 10.1038/ajg.2017.114. Epub 2017 May 2. PMID 28462914
- [Background] Buxbaum J, Quezada M, Chong B, Gupta N, Yu CY, Lane C, Da B, Leung K, Shulman I, Pandol S, Wu B. The Pancreatitis Activity Scoring System predicts clinical outcomes in acute pancreatitis: findings from a prospective cohort study. Am J Gastroenterol. 2018 May;113(5):755-764. doi: 10.1038/s41395-018-0048-1. Epub 2018 Mar 15. PMID 29545634

DOCUMENTS (1):
  • Study Protocol (2018-07-11): https://cdn.clinicaltrials.gov/large-docs/69/NCT03642769/Prot_000.pdf